CLINICAL TRIAL: NCT03387761
Title: Phase 1B Study to Assess Safety and Efficacy of Neo-Adjuvant Bladder Urothelial Carcinoma COmbination-immunotherapy (NABUCCO)
Brief Title: Neo-Adjuvant Bladder Urothelial Carcinoma COmbination-immunotherapy
Acronym: NABUCCO
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Netherlands Cancer Institute (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N17NAB; CA209-9Y4 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2017-11-24; First posted 2018-01-02 (Actual); Last update posted 2025-03-05 (Actual); Status verified 2025-03

CONDITIONS: Urothelial Carcinoma
Keywords: Urothelial cancer; Bladder cancer; Cancer; Resectable; Operable; immunotherapy; Ipilimumab; Nivolumab; Neo-Adjuvant
MeSH Terms: conditions — Carcinoma, Transitional Cell; Urinary Bladder Neoplasms; Neoplasms | interventions — Ipilimumab; Nivolumab

STUDY DESIGN:
Intervention Model Description: Multicenter, open-label phase 1b clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Cohort 1: Ipi + Nivo (Experimental): * Day 1: Ipilimumab 3 mg/kg i.v.
  * Days 22: Ipilimumab 3 mg/kg + Nivolumab 1 mg/kg i.v.
  * Day 43: Nivolumab 3 mg/kg i.v.
  Interventions: Drug: Ipilimumab; Drug: Nivolumab
- Cohort 2a: high-Ipi + low-Nivo (Experimental): * Day 1: Ipilimumab 3 mg/kg + Nivolumab 1 mg/kg i.v.
  * Days 22: Ipilimumab 3 mg/kg + Nivolumab 1 mg/kg i.v.
  * Day 43: Nivolumab 3 mg/kg i.v.
  * Radical cystectomy or nefro/ureterectomy with appropriate lymph node dissection, day 56-84
  Interventions: Drug: Ipilimumab; Drug: Nivolumab
- Cohort 2b: low-Ipi + high-Nivo (Experimental): * Day 1: Ipilimumab 1 mg/kg + Nivolumab 3 mg/kg i.v.
  * Days 22: Ipilimumab 1 mg/kg + Nivolumab 3 mg/kg i.v.
  * Day 43: Nivolumab 3 mg/kg i.v.
  * Radical cystectomy or nefro/ureterectomy with appropriate lymph node dissection, day 56-84
  Interventions: Drug: Ipilimumab; Drug: Nivolumab

INTERVENTIONS:
Drug: Ipilimumab — For Cohort 1:
  * Day 1: Ipilimumab 3 mg/kg
  * Days 22: Ipilimumab 3 mg/kg
  For Cohort 2a:
  * Day 1: Ipilimumab 3 mg/kg
  * Days 22: Ipilimumab 3 mg/kg
  For Cohort 2b:
  * Day 1: Ipilimumab 1 mg/kg
  * Days 22: Ipilimumab 1 mg/kg
  Other Names: BMS-734016; Yervoy
Drug: Nivolumab — For Cohort 1:
  * Day 22: Nivolumab 1 mg/kg
  * Day 43: Nivolumab 3 mg/kg
  For Cohort 2a:
  * Days 1 and 22: Nivolumab 1 mg/kg
  * Day 43: Nivolumab 3 mg/kg
  For Cohort 2b:
  - Days 1, 22 and 43: Nivolumab 3 mg/kg
  Other Names: BMS-936558; Opdivo

SUMMARY:
In cohort 1 of this study, we used an attenuated schedule of neoadjuvant ipilimumab and nivolumab. In the multicenter extension (cohort 2), 30 patients were randomized between two neoadjuvant treatment schemes, both based upon an attenuated schedule of neoadjuvant ipilimumab and nivolumab.Both cohorts are completed.

DETAILED DESCRIPTION:
This is an open-label phase Ib trial to evaluate three different schedules of preoperative ipilimumab and nivolumab. Urothelial cancer patients will be included that are diagnosed with either:

* cT3-4aN0M0 OR
* T1-4aN1-3M0

Cohort 1 (n=24):

* Day 1: Ipilimumab 3 mg/kg
* Days 22: Ipilimumab 3 mg/kg + Nivolumab 1 mg/kg
* Day 43: Nivolumab 3 mg/kg
* Day 56-84: Radical cystectomy or nefro/ureterectomy with appropriate lymph node dissection

Patients in cohort 2 (n=30) were randomized between cohort 2a and 2b

Cohort 2a (n=15):

* Day 1: Ipilimumab 3 mg/kg + Nivolumab 1 mg/kg
* Days 22: Ipilimumab 3 mg/kg + Nivolumab 1 mg/kg
* Day 43: Nivolumab 3 mg/kg
* Day 56-84: Radical cystectomy or nefro/ureterectomy with appropriate lymph node dissection

Cohort 2b (n=15):

* Day 1: Ipilimumab 1 mg/kg + Nivolumab 3 mg/kg
* Days 22: Ipilimumab 1 mg/kg + Nivolumab 3 mg/kg
* Day 43: Nivolumab 3 mg/kg
* Day 56-84: Radical cystectomy or nefro/ureterectomy with appropriate lymph node dissection

The primary endpoint for cohort 1 in this trial was safety. We determined the number of patients that had surgical resection <12 weeks from first infusion, as this is an endpoint that is clinically meaningful for this population. After surgery, patients attended study visits at day 8 and day 29. Their final study visit for physical examination and laboratory testing is at day 57 (+/- 7 days), which is scheduled to anticipate late-onset adverse events (particularly endocrine). After this final visit, patients were followed according to standard clinical guidelines. Tumor biopsies/material preservation were required at baseline and during surgery.

In cohort 2, we randomized patients between 2 arms. Here, the main secondary outcomes were:

* To compare the efficacy of pre-operative ipilimumab + nivolumab in cohort 1 (sequenced ipilimumab/nivolumab), versus cohort 2a (ipi 3 mg/kg and nivo 1 mg/kg) and cohort 2b (ipi 1 mg/kg and nivo 3 mg/kg). Efficacy was defined as the pCR rate at resection.
* Provide an estimate of ≥grade 3 immune-related toxicity in the ipi3/nivo1 and ipi1/nivo3 cohorts as opposed to the initial cohort (Cohort 1)

An important additional secondary endpoint is translational. The main testable hypothesis is that a significant percentage of nonresponse can be explained by immune-inhibitory processes. Absence of immune infiltrates, presence of significant numbers of regulatory T-cells and presence of significant numbers of myeloid-derived suppressor cells will be compared between responders and nonresponders. The efficacy will be defined as the percentage of pathological complete response (pCR) at cystectomy (secondary endpoint).

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide informed consent
2. Age ≥ 18 years
3. High-risk resectable urothelial cancer (upper urinary tract allowed) defined as stage III UC:

cT3-4aN0M0 OR cT1-4aN1-3M0 4. Refusal of neoadjuvant/induction cisplatin-based chemotherapy or patients in whom neoadjuvant cisplatin based therapy is not appropriate.

5. World Health Organization (WHO) performance Status 0 or 1. 6. Urothelial cancer is the dominant histology (>70%). 7. Formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks from diagnostic TUR available (or any other FFPE tumor specimens for upper tract tumors).8. Screening laboratory values must meet the following criteria: WBC ≥ 2.0x109/L, Neutrophils ≥1.0x109/L, Platelets ≥100 x109/L, Hemoglobin ≥5.5 mmol/L, GFR>30 ml/min, AST ≤ 2.5 x ULN, ALT ≤2.5 x ULN, Bilirubin ≤1.5 X ULN 9. Negative pregnancy test within 2 weeks of Day 1 Cycle 1 for female patients of childbearing potential.

10. For female patients of childbearing potential to use a highly effecting form(s) of contraception (i.e. one that results in a low failure rate [<1% per year] when used consistently and correctly) and to continue its use for 180 days after the last dose of immunotherapy Adequate contraceptive methods are: condom, sterilization, other barrier contraceptive measures preferably in combination with condoms, oral contraceptives, intra-uterine device.

Exclusion Criteria:

1. Subjects with active autoimmune disease in the past 2 years. Patients with diabetes mellitus, properly controlled hypothyroidism or hyperthyroidism, vitiligo, psoriasis or other mild skin disease can still be included.
2. Documented history of severe autoimmune disease (e.g. inflammatory bowel disease, myasthenia gravis).
3. Prior CTLA-4 or PD-1/PD-L1-targeting immunotherapy.
4. Known history of Human Immunodeficiency Virus, positive tests for Hepatitis B surface antigen or Hepatitis C ribonucleic acid (RNA), active tuberculosis, or other active infection requiring therapy at the time of inclusion.
5. Underlying medical conditions that, in the investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of adverse events
6. Medical condition requiring the use of immunosuppressive medications, with the exceptions of intranasal and inhaled corticosteroids or systemic corticosteroids at physiological doses, which are not to exceed 10 mg/day of prednisone, or an equivalent corticosteroid. Steroids as premedication for hypersensitivity reactions (eg, CT scan premedication) will be allowed.
7. Use of other investigational drugs before study drug administration
8. Malignancy, other than urothelial cancer, in the previous 2 years, with a high chance of recurrence (estimated >10%). Patients with low risk prostate cancer (defined as Stage T1/T2a, Gleason score

   ≤ 6, and PSA ≤ 10 ng/mL) who are treatment-naive and undergoing active surveillance are eligible.
9. Pregnant and lactating female patients.
10. Major surgical procedure within 4 weeks prior to enrolment or anticipation of need for a major surgical procedure during the course of the study other than for diagnosis.
11. Severe infections within 4 weeks prior to enrolment in the study including but not limited to hospitalization for complications of infection, bacteraemia, or severe pneumonia.
12. Significant cardiovascular disease, such as New York Heart Association cardiac disease (Class II or greater), myocardial infarction within 3 months prior to enrolment, unstable arrhythmias, or unstable angina.
13. Previous intravenous chemotherapy for bladder cancer. Prior chemoradiation is allowed.
14. Patients in whom use of a colon segment for urinary diversion is planned

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2025-01-07 (Actual)

PRIMARY OUTCOMES:
Number of patients that had surgical resection <12 weeks after study start (Cohort 1) | At 12 weeks
  Percentage of patients that underwent surgery within 12 weeks after study start were assessed

SECONDARY OUTCOMES:
Efficacy of immunotherapy, assessed by by the percentage of pathological complete response rate (pCR) after cystectomy (Cohort 1, followed by Cohort 2a versus 2b) | At 12 weeks
  pCR rate after cystectomy according to pathological response criteria
Differences in immune infiltrates in responders vs nonresponders | At 12 weeks
  Resistance mechanisms are explored by comparing immune (cell) infiltrates in responders and nonresponders in pre- and post treatment tissue [Multiplex immunohistochemistry, RNA seq]
T-cell (dys)functionality as measured by comparing the transcriptome of tumor-specific T cells in intra-patient pre- and post therapy tissue | At 12 weeks
  This component is done in a minority of patients on T cell lysates if a re-TUR (transurethral resection) pre-treatment was done.
Explore whether radiomics-based predictive models can be established for immunotherapy responders vs non-responders (Cohort 1) | At 12 weeks
  CT and MRI images will be assessed in this manner to optimize recognition of an immunotherapy response.
Provide an estimate of ≥grade 3 immune-related toxicity in cohorts 2a versus 2b | At 12 weeks
  Immune-related toxicity were compared between cohhort 1 and cohort 2 and between cohorts 2a and 2b
Monitor peri-surgical complications. | Until 90 days after surgery.
  peri-operative complications and morbidity were graded according to the Clavien-Dindo classification.
ctDNA in plasma during follow-up | During follow-up and with disease recurrence
  Assessment of ctDNA in plasma during follow-up and at recurrence
As part of regular follow-up after radical surgery, follow-up CT scans were made after 1 and 2 years. | Until 2 years after surgery (not part of primary study assessment)
  As part of regular follow-up after radical surgery, follow-up CT scans were made after 1 and 2 years. Additional scans were performed according to local standards.

CONTACTS AND LOCATIONS:
Overall Officials: Michiel MS van der Heijden, Dr., Principal Investigator — NKI-AvL
Locations (3):
- Netherlands (3):
  - Antoni van Leeuwenhoek ziekenhuis, Amsterdam, North Holland
  - Radboud UMC, Nijmegen
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Stockem CF, van Dorp J, van Dijk N, Vis DJ, Harkes R, van den Broek B, Alkemade M, Broeks A, Hendricksen K, Boellaard TN, de Feijter JM, van Montfoort ML, Daletzakis A, van der Heijden AG, Meijer RP, Mehra N, Wessels LFA, van Rhijn BWG, Suelmann BBM, van der Heijden MS. Final clinical analysis of pre-operative ipilimumab and nivolumab in locally advanced urothelial cancer and exploration of tumor-draining lymph node composition: The NABUCCO trial. Eur J Cancer. 2025 Oct 16;229:115731. doi: 10.1016/j.ejca.2025.115731. Epub 2025 Aug 21. PMID 40934711
- [Derived] van Dorp J, Pipinikas C, Suelmann BBM, Mehra N, van Dijk N, Marsico G, van Montfoort ML, Hackinger S, Braaf LM, Amarante T, van Steenis C, McLay K, Daletzakis A, van den Broek D, van de Kamp MW, Hendricksen K, de Feijter JM, Boellaard TN, Meijer RP, van der Heijden AG, Rosenfeld N, van Rhijn BWG, Jones G, van der Heijden MS. High- or low-dose preoperative ipilimumab plus nivolumab in stage III urothelial cancer: the phase 1B NABUCCO trial. Nat Med. 2023 Mar;29(3):588-592. doi: 10.1038/s41591-022-02199-y. Epub 2023 Feb 2. PMID 36732628
- [Derived] van Dijk N, Gil-Jimenez A, Silina K, Hendricksen K, Smit LA, de Feijter JM, van Montfoort ML, van Rooijen C, Peters D, Broeks A, van der Poel HG, Bruining A, Lubeck Y, Sikorska K, Boellaard TN, Kvistborg P, Vis DJ, Hooijberg E, Schumacher TN, van den Broek M, Wessels LFA, Blank CU, van Rhijn BW, van der Heijden MS. Preoperative ipilimumab plus nivolumab in locoregionally advanced urothelial cancer: the NABUCCO trial. Nat Med. 2020 Dec;26(12):1839-1844. doi: 10.1038/s41591-020-1085-z. Epub 2020 Oct 12. PMID 33046870